CLINICAL TRIAL: NCT03550820
Title: Energy Metabolism for the Patients With Pulmonary Mycobacterium Avium Complex
Status: Completed | Type: Observational
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 28-2
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary MAC; Energy Metabolism; Emaciation
Keywords: pulmonary MAC; energy metabolism
MeSH Terms: conditions — Emaciation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aim to examine energy metabolism in patients with pulmonary MAC and clarify the causes of emaciation. We will also investigate the following: the relation between energy metabolism and degree of pulmonary MAC progression; relations among hospitalization, mortality rate, and time-course of changes in energy metabolism; and factors that affect energy metabolism.

DETAILED DESCRIPTION:
Patients with pulmonary MAC with a lower BMI than healthy individuals also have a significantly poorer prognosis than those of normal weight. Emaciation in such patients is thought to be caused by destruction of lung structure from disease progression and an increased resting metabolic rate caused by the increased load from breathing; however, causes of emaciation and details of energy metabolism in these patients have not been studied.

Elucidating details of energy metabolism and causes of emaciation in patients with pulmonary MAC could provide the basis for improvement in nutritional status and activities of daily living through early nutrition therapy and rehabilitation. We propose to clarify the following:

Energy metabolism in patients with pulmonary MAC, including resting metabolic rate, calorie intake and consumption, and hormonal secretions.

Relation between energy metabolism and degree of pulmonary MAC progression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pulmonary MAC.

Exclusion Criteria:

* Subjects with severe cardiovascular disease, diabetes, neurological disease, renal failure, endocrine disease and malignant neoplasm.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Petients with pulmonary MAC
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Relation between energy balance and pulmonary MAC severity | Three years

SECONDARY OUTCOMES:
Relation between inflammation (CRP et.) and pulmonary MAC severity | Three years
Relation between bone mineral density and pulmonary MAC severity | Three years
Relation between hormone secretion and pulmonary MAC severity | Three years
Relation between pulmonary function and pulmonary MAC severity | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan